CLINICAL TRIAL: NCT05912816
Title: Perioperative Disitamab Vedotin and Tislelizumab Followed by Nephron-Sparing Surgery in High-Risk Upper Tract Urothelial Carcinoma: A Phase 2 Trial (DISTINCT-I)
Brief Title: Combination of DV and Tislelizumab for Renal Preservation in High-risk UTUC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Tianjin Medical University Second Hospital (Other); Peking University First Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DISTINCT-I
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma; Kidney Preservation; HER-2 ADC; PD-1antibody
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: In this trial, RC48 was scheduled to be administered at a dose of 2.0 mg/kg every 3 weeks, with the first dose on day 1 of the first cycle.
  Tislelizumab was administered at a dose of 200 mg every 3 weeks, with the first dose on day 1 of the first 21-day cycle. The drug is diluted with normal saline and administered by intravenous drip for one hour.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 Combined With Tislelizumab (Experimental): In this trial, RC48 was scheduled to be administered at a dose of 2.0 mg/kg every 3 weeks, with the first dose on day 1 of the first cycle.
  Tislelizumab was administered at a dose of 200 mg every 3 weeks, with the first dose on day 1 of the first 21-day cycle. The drug is diluted with normal saline and administered by intravenous drip for one hour.
  Interventions: Drug: RC48 Combined With Tislelizumab

INTERVENTIONS:
Drug: RC48 Combined With Tislelizumab — In this trial, RC48 was scheduled to be administered at a dose of 2.0 mg/kg every 3 weeks, with the first dose on day 1 of the first cycle.
  Tislelizumab was administered at a dose of 200 mg every 3 weeks, with the first dose on day 1 of the first 21-day cycle. The drug is diluted with normal saline and administered by intravenous drip for one hour.

SUMMARY:
This is a prospective, open, multiple-center clinical study of renal preservation therapy in high-risk upper urinary tract urothelial carcinoma patients . The study was conducted in accordance with the Good Practice for Quality Control of Clinical Trials for Pharmaceutical Products (GCP). Approximately 20 subjects will be enrolled to evaluate the efficacy and safety of RC48 (2.0 mg/kg intravenously every 3 weeks) combined with Tislelizumab (200mg intravenously every 3 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. ECOG 0~2;
2. HER-2 IHC 0-3+;
3. Subjects underwent cystoscopic/ureteroscopic biopsy, exfoliation cytology, and CT/MRI diagnosis;
4. Patients were judged to be high-risk urothelial carcinoma of the upper urinary tract (meeting any of the following risk factors: hydronephrosis, tumor diameter ≥2cm, high-grade, multiple tumors in cytology, previous history of radical cystectomy for high-grade bladder cancer, biopsy pathology with other tissue components);
5. High-risk UTUC(excluding low-risk UTUC),including renal pelvic tumors (cT1-T3, N0) or ureteral tumors (cT1-T3, N0-N1) M0;
6. Patients with indications of absolute or relative renal protection (only kidney, renal insufficiency: eGFR < 60 ml/min)
7. Have the desire to protect the kidney;
8. There is no indication of absolute or relative kidney preservation, but patients have a strong desire to preserve kidney.
9. Has and agrees to provide cystoscopic/ureteroscopic biopsy tissue specimens and to reserve pre-treatment blood,
10. Urine and biopsied biological samples;
11. Predicted survival ≥3 months;
12. Major organ function is normal (14 days prior to enrollment)
13. International Normalized ratio (INR), activated partial thromboplastin time (aPTT) : ≤1.5× ULN (This criterion only applies to patients who are not receiving anticoagulant therapy; Patients receiving anticoagulant therapy should keep anticoagulants within therapeutic limits);
14. Did not receive systemic corticosteroid medication within 4 weeks prior to treatment;
15. Fertile men or women who are at risk of becoming pregnant must use a highly effective contraceptive method during the trial (such as oral contraceptives, intrauterine devices, controlled sexual desire or barrier contraception combined with spermicide) and continue using contraception for 12 months after the end of treatment;
16. The subjects voluntarily joined the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Previously received anti-PD-1, anti-PD-L1, anti-PD-L2 therapy, including adjuvant therapy stage;
2. Known allergy to recombinant humanized anti-PD-1 monoclonal antibody drugs and their components;
3. Had received other antitumor therapy (including corticosteroid therapy, immunotherapy) or participated in other clinical studies within 4 weeks prior to the study treatment, or had not recovered from the previous toxicity (except for 2 degrees of hair loss and 1 degree of neurotoxicity);
4. Pregnant or lactating women;
5. Positive HIV test result;
6. People with active hepatitis B or C
7. HBsAg or HBcAb positive patients also detected HBV DNA copy number positive (quantitative detection limit is 500IU/ml, or reach the positive value of the study center); Screening studies of such patients must test for HBV DNA;
8. Patients who tested positive for HCV antibodies were enrolled in this study only if the PCR results of HCV RNA were negative.
9. A clear history of active tuberculosis;
10. Have active autoimmune diseases that have required systemic treatment within the past 2 years (e.g., with disease-regulating drugs, corticosteroids, or immunosuppressive drugs) that allow for relevant replacement therapy (e.g., thyroxine, pancreatic hormone, or physiologic corticosteroid replacement therapy for renal or pituitary insufficiency);
11. Other serious, uncontrolled concomitant diseases that may affect protocol adherence or interfere with interpretation of results, These include active opportunistic or progressive (severe) infections, uncontrolled diabetes, cardiovascular disease (heart failure of Grade Ⅲ or Ⅳ as defined by the New York Heart Association scale, heart block above grade Ⅱ, myocardial infarction within the past 6 months, unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc.) Or pulmonary disease (history of interstitial pneumonia, obstructive pulmonary disease, and symptomatic bronchospasm);
12. Received live vaccine within 4 weeks prior to the start of treatment;
13. Have previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
14. Major surgical procedures (excluding diagnostic surgery) within 4 weeks prior to the start of treatment; Those who have a history of psychotropic drug abuse and cannot abstain or have a history of mental disorders;
15. A large amount of pleural effusion or ascites accompanied by clinical symptoms or requiring symptomatic treatment;
16. Have had other unhealed malignancies in the past 5 years, excluding those that are apparently cured or curable, such as basal or squamous cell skin cancer, localized low-risk prostate cancer, carcinoma in situ of the cervix or carcinoma in situ of the breast; Remarks: Patients with localized low-risk prostate cancer (defined as stage ≤T2a, Gleason score ≤6, and PSA≤10ng/mL at the time of prostate cancer diagnosis (as measured) who had received radical therapy and had no biochemical recurrence of prostate specific antigen (PSA) were eligible to participate in this study);
17. Bladder cancer (MIBC);
18. Other severe, acute, or chronic medical or psychiatric conditions or laboratory abnormalities that, according to the investigator, may increase the risks associated with study participation or may interfere with the interpretation of the study results.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2025-11-03 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
kidney-intact event-free survival (KI-EFS) | up to 1 year
  the time from enrollment to any event, including high-risk UTUC local recurrence(tumor size ≥2 cm, local invasion on CT or MRI, hydronephrosis, or multifocality), distant metastasis, death from any cause, or conversion to RNU

SECONDARY OUTCOMES:
clinical complete response | 3 month before surgery
  The rate of CCR is defined by negative ureteroscope, urine cytology, and negative imaging
clinical complete response | 4 month after surgery
  The rate of CCR is defined by negative ureteroscope, urine cytology, and negative imaging
disease-free survival | up to 2 year
  the time from enrollment to any disease recurrence (excluding isolated bladder recurrence) or death from any cause
the proportion of adverse events | up to 2 year
  adverse events graded according to CTCAE version 5.0
the proportion of RUN | up to 2 year
  The proportion of patients undergoing radical surgery for UTUC (upper tract urothelial carcinoma) after enrollment.
renal function preservation | up to 1 year
  the change in eGFR from baseline to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ethics Committee of Shanghai Renji Hospital, Shanghai, Shanghai Municipality, China